CLINICAL TRIAL: NCT02388789
Title: Effects of Changes in Foot Skin Temperature on Plantar-surface Mechanoreceptor Sensitivity and Balance Control
Brief Title: Foot Skin Temperature and Balance Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Stephen Perry (Other)
Responsible Party: Sponsor-Investigator, Dr. Stephen Perry, Professor, Wilfrid Laurier University
Organization: Wilfrid Laurier University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KB_CMTS
Record Dates: First submitted 2015-02-28; First posted 2015-03-17 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Mechanoreceptor; Perpherial Hypothermia
Keywords: sensory receptors; balance control; gait; temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active movement (Experimental): use a light treadmill run to raise feet temperature
  Interventions: Other: active movement

INTERVENTIONS:
Other: active movement — same as arm description

SUMMARY:
The purpose of this study is to investigate whether mechanoreceptor sensitivity of the sole of the feet increases with increased foot temperature and how a heightened sensation may improve characteristics of balance control and gait. As an extension, the investigators also want to determine whether lower limb movement is an efficient activity of increasing foot temperature. There are several objectives of this study. The investigators want to determine the effect of active recovery (via lower limb movements) on increasing plantar temperature, determine the effect of increased plantar temperature on plantar sensation and determine the effect of increased plantar sensation on balance control and gait characteristics. Participants will be asked to complete various tasks under different conditions. Conditions include decreased feet temperature via ice bath emersion, baseline feet temperature (participant's normal temperature after a ten minute equilibration period), and increased feet temperature via active movement of the lower limb. Tasks include walking across the room, performing active movement of the lower limb and a 10 minute treadmill walk. Gait movement will be collected with a three-dimensional motion capture system (Optotrak) and force plates. Feet temperature and sensation information will be collected with a temperature probe (infrared) and monofilaments.

DETAILED DESCRIPTION:
Between 10-15 healthy young adults of both males and females will be recruited. A screening questionnaire will be administered to ensure that participants are appropriate for the study.

Upon arrival, participants will be required to sit with their feet slightly elevated from the ground, resting on a stool for 10 minutes to allow for adjustment to room temperature (equilibration). During this time, participants will complete a questionnaire regarding their experiences with the temperature of their feet including questions similar to, "On average would you say that you have cold feet, average feet or warm feet? Describe your feet's ability to adapt to temperature changes. Do you experience a tingling feeling on the bottom of your feet?" Following the equilibration period, the researcher will place 12 infrared markers on the participant. The participant will then receive a brief outline of the procedure and appropriate instructions before beginning the experiment.

All trials will be performed barefoot. There will be a total of 3 types of testing. The first is a monofilament test. The researcher will apply varying monofilaments sizes to the participants' soles of their feet. These test are included to measure touch sensation of the sole of the foot. The second is a One Leg Stance Test where the participant will stand on a force plate, balanced on one leg for 30 seconds per trial while Optotrak information is collected. The participant will complete a total of 3 trials. The third is the Gait Termination Test where the participant will be instructed to walk along 6 metres over 2 force plates. A total of 10 trials will be completed with 3 randomized trials where the participant will be instructed to terminate their gait unexpectedly (by a buzzer) before reaching the force plates. Optotrak information will be collected simultaneously. The researcher will record plantar temperature intermittently in between the above tests and different conditions. The infrared temperature probe does not make any contact with the skin.

The specific outline of the procedure including the order of the conditions and tasks are explained here. The first condition is the Baseline Condition where all 3 types of tests will be administered. Then the participant's feet will be immersed in an ice bath at 2-3 degrees Celsius for 10-15 minutes (with their feet temperature recorded every 2 minutes) in preparation for the Decreased Feet Temperature Condition. Here, all 3 types of tests will be administered. Then each participant will actively recover by walking on a treadmill at a speed of 3.5 miles/hour and grade of 0% for 10 minutes, to prepare the for Increased Feet Temperature Condition. Intermittent foot temperature measurements will be taken every 2 minutes during the treadmill walk. After the 10 minute walk, all 3 types of tests will be administered. This will be the end of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years of age

Exclusion Criteria:

* CONDITIONS AFFECTING BALANCE,
* CONDITIONS AFFECTING CIRCULATION (EX: FROSTBITE), AND
* ANY OTHER CONDITIONS AFFECT SENSORY PERCEPTION.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Balance stability margin (how close their body gets to perimeter of their base of support) | within subject (every 40 minutes over 2 hours), same day
  change in ability to control body movements during standing and walking

SECONDARY OUTCOMES:
Sensory threshold (change in perception of touch pressure on the sole of the foot, taken after every change in foot temperature) | within subject (every 40 minutes over 2 hours), same day
  change in perception of touch pressure on the sole of the foot, taken after every change in foot temperature
Foot skin temperature | within subject (every 40 minutes over 2 hours), same day
  change in infrared measurement of skin temperature

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Perry, PhD, Study Director — Wilfrid Laurier University
Locations (1):
- WLU Biomechanics Laboratory, Waterloo, Ontario, Canada